CLINICAL TRIAL: NCT00709384
Title: Prevention of Atrial Tachycardia After a Right Atriotomy II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Peter Lukac, MD, PhD, Skejby Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030198B
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prophylactic intervention (Experimental): We performed a prophylactic peroperative linear lesions connecting the tricuspid annulus with a right atriotomy (surgical dissection plus cryoablation) and the atriotomy with the inferior caval vein (cryoablation alone). Conduction times between electrodes placed on both sides of the lesions are measured on the second postoperative day. Coronary angiography and electrophysiology study using an electroanatomic mapping system to assess conduction across the line and to try to induce atrial flutter are performed three month after the operation.
  There is only an intervention arm, no control arm
  Interventions: Procedure: Prophylactic surgical lesion

INTERVENTIONS:
Procedure: Prophylactic surgical lesion — A prophylactic peroperative linear lesions connecting the tricuspid annulus with a right atriotomy (surgical dissection plus cryoablation) and the atriotomy with the inferior caval vein (cryoablation alone).

SUMMARY:
The investigators performed a prophylactic peroperative linear lesions connecting the tricuspid annulus with a right atriotomy and the atriotomy with the inferior caval vein to prevent atrial flutter on 15 consecutive adult patients undergoing surgery for congenital heart disease. Conduction time between electrodes placed on both sides of the lesions is measured on the second postoperative day. Coronary angiography and electrophysiology study using an electroanatomic mapping system to assess conduction across the line are performed three month after the operation.

DETAILED DESCRIPTION:
We perform a prophylactic peroperative linear lesions connecting the tricuspid annulus with a right atriotomy (surgical dissection plus cryoablation) and the atriotomy with the inferior caval vein (cryoablation alone) to prevent atrial flutter on 15 consecutive adult patients undergoing surgery for congenital heart disease. Conduction times between electrodes placed on both sides of the lesions are measured on the second postoperative day. Coronary angiography and electrophysiology study using an electroanatomic mapping system to assess conduction across the line and to try to induce atrial flutter are performed three month after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for corrective operation for congenital heart disease with the use of a right lateral atriotomy,
2. Age >18 years,
3. Ability to give an informed consent.

Exclusion Criteria:

1. Acute operation
2. Chronic atrial fibrillation
3. Indication for MAZE procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
completeness of the lines of block | 3 month

SECONDARY OUTCOMES:
safety | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Skejby Hospital, Aarhus, Denmark